CLINICAL TRIAL: NCT05655533
Title: Added Value of Diffusion Weighted MRI in Evaluation of Sacroiliitis in Newly Diagnosed Patients of Spondyloarthropathy.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lamia a Arafat, Resident Physician, Assiut University
Other Study IDs: 455457
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Spondyloarthropathy and Sacroilitis
MeSH Terms: conditions — Spondylarthropathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients who clinically suspected to have early spondyloarthropathy: Adult patients who clinically suspected to have early spondyloarthropathy in acute stage.
  At least 4 of 5 criteria for inflammatory low back pain have to be fulfilled
  Interventions: Diagnostic Test: Magnetic resonance Imaging scanners of sacroiliac joints.

INTERVENTIONS:
Diagnostic Test: Magnetic resonance Imaging scanners of sacroiliac joints. — Patients will undergo MR imaging examinations with a closed 1.5-Tesla Magnetic resonance Imaging scanners of sacroiliac joints.
  The patients will be imaged in the supine position using a body phased-array coil.
  Evaluate the added value of DWI in detection of acute sacroiliitis and whether ADC values can be helpful in detection and differentiation of active stage, so determine whether supplementation of DWI with quantitative ADC mapping to the routine MR examination is of great value as non-invasive tool or not

SUMMARY:
Spondyloarthropathy encompasses a group of chronic immune-mediated rheumatic inflammatory diseases characterized by axial joint inflammation, peripheral arthritis, enthesitis, dactylitis and extra-articular features.

Axial spondyloarthritis (SpA) has significant social and psychiatric impacts [2, 3] and affects quality-of-life (4-5).Early disease diagnosis is becoming more important as it will facilitate early therapeutic interventions (6).

There's no "gold standard" feature for diagnosing axSpA. It's diagnosed through a combination of patient history, clinical examination, laboratory findings a and imaging tests, such as X-ray and MRI.

Sacroiliitis is commonly the first manifestation and an important indicator of the diagnosis and classification of the the disease. (7) Radiographic sacroiliitis is a key criterion. However, sole reliance on radiographs is associated with significant diagnostic delay [8]. Magnetic Resonance Imaging (MRI) can detect axial inflammation before radiographic changes.

Diffusion-weighted imaging (DWI) offers a new approach to assess inflammation. Recently several studies have shown that DWI is an effective tool in early diagnosis of axSpA (14-16). Furthermore, the ADC value may serve as a quantitative biomarker of disease activity, allowing monitoring and guiding treatment. (17-18)

DETAILED DESCRIPTION:
Spondyloarthropathy encompasses a group of chronic immune-mediated rheumatic inflammatory diseases characterized by axial joint inflammation, peripheral arthritis, enthesitis, dactylitis and extra-articular features such as psoriasis, uveitis, inflammatory bowel disease (crohns and ulcerative colitis) [1].

Axial spondyloarthritis (SpA) has significant social and psychiatric impacts [2, 3] and affects quality-of-life (4-5). Patients often experience prolonged delays in diagnosis. Early disease diagnosis is becoming more important as it will facilitate early therapeutic interventions (6).

There's no "gold standard" feature for diagnosing axSpA. It's diagnosed through a combination of patient history, clinical examination, laboratory findings as blood tests (both for HLA-B27 and for markers of inflammation, such as C-reactive protein), and imaging tests, such as X-ray and MRI.

Sacroiliitis is commonly the first manifestation and an important indicator of the diagnosis and classification of the the disease. (7) Radiographic sacroiliitis is a key criterion. However, sole reliance on radiographs is associated with significant diagnostic delay [8]. Magnetic Resonance Imaging (MRI) can detect axial inflammation before radiographic changes. (9) So with the development of Assessment of Spondyloarthritis International Society (ASAS) classification criteria for ax-SpA, MRI is increasingly being used to early diagnose and monitor disease activity. (10) Diffusion-weighted imaging (DWI) offers a new approach to assess inflammation. It is a functional MRI technique that can non-invasively asses the random movements of water molecules through the measurements of the ADC value. (11). Inflammation produces an increase in the apparent diffusion coefficient (ADC) of water molecules in affected tissues, probably owing to an increase in the ratio of extracellular to intracellular water. (12-13) Recently several studies have shown that DWI is an effective tool in early diagnosis of axSpA (14-16). Furthermore, the ADC value may serve as a quantitative biomarker of disease activity, allowing monitoring and guiding treatment. (17-18)

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who are suspected clinically to have early spondyloarthropathy with acute sacroiliitis.

Exclusion Criteria:

* Known patients with chronic spondyloarthropathy under medical treatment.
* Patients with previous surgical operations and metallic screws fixation at pelvic region.
* Patients refused the examination.
* Patients with contraindication to MRI as claustrophobia, pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients who clinically suspected to have early spondyloarthropathy in acute stage, referred from rheumatologists or orthopedic clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-12-10 (Estimated); Primary Completion 2024-05-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
value of diffusion weighted MRI in evaluation of sacroiliitis in newly diagnosed patients of spondyloarthropathy. | one year
  Diagnostic value of Diffusion weighted MRI of Sacroiliac joint compared to Conventional sequence MRI of sacroiliac joint for the diagnosis of sacroiliitis.

SECONDARY OUTCOMES:
Early diagnosis of spondyloarthropathy | one year
  Early diagnosis of spondyloarthropathy by early detection of sacroiliitis in clinically suspected patients will facilitate early therapeutic interventions thus lead to dramatic improvements in the management of axial SpA by reducing symptoms and preserving functional status.

REFERENCES:
- [Background] Sieper J, Poddubnyy D. Axial spondyloarthritis. Lancet. 2017 Jul 1;390(10089):73-84. doi: 10.1016/S0140-6736(16)31591-4. Epub 2017 Jan 20. PMID 28110981
- [Background] Chan CYY, Tsang HHL, Lau CS, Chung HY. Prevalence of depressive and anxiety disorders and validation of the Hospital Anxiety and Depression Scale as a screening tool in axial spondyloarthritis patients. Int J Rheum Dis. 2017 Mar;20(3):317-325. doi: 10.1111/1756-185X.12456. Epub 2014 Oct 7. PMID 25293872
- [Background] Zink A, Braun J, Listing J, Wollenhaupt J. Disability and handicap in rheumatoid arthritis and ankylosing spondylitis--results from the German rheumatological database. German Collaborative Arthritis Centers. J Rheumatol. 2000 Mar;27(3):613-22. PMID 10743798
- [Background] Ward MM. Health-related quality of life in ankylosing spondylitis: a survey of 175 patients. Arthritis Care Res. 1999 Aug;12(4):247-55. PMID 10689989
- [Background] Chan CWS, Tsang HHL, Li PH, Lee KH, Lau CS, Wong PYS, Chung HY. Diffusion-weighted imaging versus short tau inversion recovery sequence: Usefulness in detection of active sacroiliitis and early diagnosis of axial spondyloarthritis. PLoS One. 2018 Aug 7;13(8):e0201040. doi: 10.1371/journal.pone.0201040. eCollection 2018. PMID 30086145
- [Background] Lambert RG, Bakker PA, van der Heijde D, Weber U, Rudwaleit M, Hermann KG, Sieper J, Baraliakos X, Bennett A, Braun J, Burgos-Vargas R, Dougados M, Pedersen SJ, Jurik AG, Maksymowych WP, Marzo-Ortega H, Ostergaard M, Poddubnyy D, Reijnierse M, van den Bosch F, van der Horst-Bruinsma I, Landewe R. Defining active sacroiliitis on MRI for classification of axial spondyloarthritis: update by the ASAS MRI working group. Ann Rheum Dis. 2016 Nov;75(11):1958-1963. doi: 10.1136/annrheumdis-2015-208642. Epub 2016 Jan 14. PMID 26768408
- [Background] Rudwaleit M, van der Heijde D, Khan MA, Braun J, Sieper J. How to diagnose axial spondyloarthritis early. Ann Rheum Dis. 2004 May;63(5):535-43. doi: 10.1136/ard.2003.011247. PMID 15082484
- [Background] Bozgeyik Z, Ozgocmen S, Kocakoc E. Role of diffusion-weighted MRI in the detection of early active sacroiliitis. AJR Am J Roentgenol. 2008 Oct;191(4):980-6. doi: 10.2214/AJR.07.3865. PMID 18806131
- [Background] Carmona R, Harish S, Linda DD, Ioannidis G, Matsos M, Khalidi NA. MR imaging of the spine and sacroiliac joints for spondyloarthritis: influence on clinical diagnostic confidence and patient management. Radiology. 2013 Oct;269(1):208-15. doi: 10.1148/radiol.13121675. Epub 2013 Jun 27. PMID 23813394
- [Background] Khoo MM, Tyler PA, Saifuddin A, Padhani AR. Diffusion-weighted imaging (DWI) in musculoskeletal MRI: a critical review. Skeletal Radiol. 2011 Jun;40(6):665-81. doi: 10.1007/s00256-011-1106-6. Epub 2011 Feb 12. PMID 21311884